CLINICAL TRIAL: NCT03221582
Title: Impact of HCV Therapy on Cardiovascular Risk and Bone Health
Brief Title: Impact of Hepatitis C Therapy and Bone Health
Acronym: HCV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Site unable to recruit the agreed upon number of participants
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISP 54850
Record Dates: First submitted 2017-06-27; First posted 2017-07-18 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Human Immunodeficiency Virus; Hepatitis C
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EBR/GZR (Zepatier) - HCV/HIV co-infected (Experimental): Drug: Elbasvir (EBR) 50 mg and Grazoprevir (GZR) 100 mg single tablet by mouth, once daily.
  Interventions: Drug: EBR/GZR
- EBR/GZR (Zepatier) - HCV monoinfected (Experimental): Drug: Elbasvir (EBR) 50 mg and Grazoprevir (GZR) 100 mg single tablet by mouth, once daily.
  Interventions: Drug: EBR/GZR

INTERVENTIONS:
Drug: EBR/GZR — Elbasvir and Grazoprevir (EBR/GZR) tablet by mouth, once daily.
  Other Names: Zepatier

SUMMARY:
An evaluation of the impact of Elbasvir and Grazoprevir (EBR/GZR) HCV therapy on the heart risk and bone health of HCV mono-infected and HIV/HCV co-infected patients.

DETAILED DESCRIPTION:
Both HCV and HIV are associated with an increased risk of osteoporosis and osteoporotic fractures among HIV-infected patients and the general population. While HIV significantly increases cardiovascular risk, the contribution of HCV to cardiovascular disease (CVD) is less certain. Increased inflammation could potentially underlie the effect of HCV on CVD, bone health, and other extra-hepatic complications. HCV appears to remain an independent predictor of osteoporotic fractures even after controlling for severity of liver disease. The impact of HCV therapy on inflammation, CVD and bone health is unclear. Our previous studies suggest a beneficial impact of interferon therapy on bone turnover and some CVD markers, while others studies have found on-treatment increases in bone mineral density with interferon-based therapy. Whether these are related to the interferon itself or the virologic response, and whether changes in biomarkers lead to improved fracture risk or CVD morbidity is uncertain. Investigator propose to conduct a prospective analysis of markers of inflammation, immune activation, and bone turnover as well as bone mineral density (BMD) among both HIV/HCV co-infected and HCV mono-infected patients undergoing treatment with the novel direct-acting antiviral elbasvir/grazoprevir (EBR/GZR). Should EBR/GZR therapy significantly improve CV risk and bone health, it would be an additional benefit and indication for its use in HCV therapy.

ELIGIBILITY:
Inclusion Criteria:

1. HCV antibody and HCV RNA positive
2. HCV Genotype 1a, 1b, or 4
3. Liver staging assessment:

   a. Cirrhosis will be defined by any of the following: i. A liver biopsy prior to day 1 of this study showing cirrhosis (F4) ii. Fibroscan within 12 calendar months of day 1 of this study showing cirrhosis with result > 12.5 kPa iii. FibroSURE performed during screening with a score > 0.75 and APRI > 2 b. Absence of cirrhosis will be defined by any of the following: i. Liver biopsy performed within 24 months of day 1 of this study showing absence of cirrhosis ii. Fibroscan performed within 12 months of day 1 of this study with a result of ≤ 12.5 kPa iii. FibroSURE score ≤ 0.48 and APRI ≤ 1 during screening
4. If HIV co-infected, HAART regimen will consist of two NRTIs (abacavir, tenofovir disoproxil fumarate or tenofovir alafenamide, each in combination with lamivudine or emtricitabine) with one of the following 3rd agents:

   1. raltegravir
   2. dolutegravir
   3. rilpivirine HIV co-infected patients must be on their stable HAART regimen for at least 6 months, with HIV viral load < 50 c/mL at screening

Exclusion Criteria:

1. Hepatitis B surface antigen positivity
2. Decompensated cirrhosis (Child Pugh B or C)
3. Any prior hepatitis C treatment
4. Pregnant or nursing
5. Treatment with any medication specifically contraindicated with EBR/GZR or not recommended for concomitant use as per the prescribing label (Table 2)
6. Age less than 18
7. Prisoners or subjects otherwise involuntarily incarcerated
8. Absence of signed informed consent by patient or appropriate surrogate
9. Known hypersensitivity to elbasvir or grazoprevir
10. For patients with genotype 1a, one more of the following mutations on baseline NS5A genotype: M28, Q30, L31, or Y93

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HCV mono-infected patients and HIV/HCV co-infected patients | 48 weeks
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, positron emission tomography (PET) scanning for arterial inflammation, coronary calcification and myocardial viability.

SECONDARY OUTCOMES:
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HCV mono-infected patients. | Biomarkers of inflammation and bone turnover measured at week 0 of therapy.
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by dual energy x-ray absorptiometry (DXA) scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HCV mono-infected patients. | Bone mineral density measured at week 0 of therapy
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HCV mono-infected patients. | Biomarkers of inflammation and bone turnover measured at week 12 of therapy.
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HCV mono-infected patients. | Biomarkers of inflammation and bone turnover measured at week 24 of therapy.
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HCV mono-infected patients. | Bone mineral density measured at week 48 of therapy.
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HIV/HCV co-infected patients. | Biomarkers of inflammation and bone turnover measured at week 0 of therapy.
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HIV/HCV co-infected patients. | Bone mineral density measured at week 0 of therapy
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HIV/HCV co-infected patients. | Biomarkers of inflammation and bone turnover measured at week 12 of therapy.
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HIV/HCV co-infected patients. | Biomarkers of inflammation and bone turnover measured at week 24 of therapy.
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).
Impact of EBR/GZR HCV therapy on the cardiovascular risk and bone health of HIV/HCV co-infected patients. | Biomarkers of inflammation and bone turnover measured at week 48 of therapy.
  Cardiovascular health will be assessed by serologic markers of inflammation; in addition to, PET scanning for arterial inflammation, coronary calcification and myocardial viability. Bone health will be assessed by serological markers of bone turnover and bone mineral density (BMD) by DXA scan and trabecular bone score (TBS).

CONTACTS AND LOCATIONS:
Overall Officials: Roger Bedimo, MD, Principal Investigator — Dallas VAMC
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No